CLINICAL TRIAL: NCT04527757
Title: Duration of Inhalation Versus Intravenous Anaesthesia Induction in Paediatric Patients: Prospective Observational Trial
Brief Title: Duration of Anaesthesia Induction in Paediatric Patients: Prospective Observational Trial
Acronym: Induration
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, prof.MD,Ph.D., Brno University Hospital
Other Study IDs: KDAR FN Brno 2020/09
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anaesthesia Induction
Keywords: Anaesthesia; Paediatric; Inhalation; Intravenous
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric patients with inhalation induction: The measurement will begin after the patient's arrival at the operating theatre, after the control of the documentation and beginning of the vital signs monitoring. The measurement will be terminated at the occurence of the first ETCO2 wave, after securing the airway with laryngeal mask or orotracheal intubation. For the inhalation induction sevoflurane will be used (in the mixture with O2 + air, or O2 + N2O).
  Interventions: Procedure: Inhalation induction
- Paediatric patients with intravenous induction: The measurement will begin after the patient's arrival at the operating theatre, after the control of the documentation and beginning of the vital signs monitoring. The measurement will be terminated at the occurence of the first ETCO2 wave, after securing the airway with laryngeal mask or orotracheal intubation. For the inhalation induction sevoflurane will be used (in the mixture with O2 + air, or O2 + N2O). For the intravenous induction, commonly used induction anaesthetics will be used (propofol, etomidate, ketamine, midazolam).
  Interventions: Procedure: Intravenous induction

INTERVENTIONS:
Procedure: Inhalation induction — For the inhalation induction sevoflurane will be used (in the mixture with O2 + air, or O2 + N2O).
  Other Names: Anaesthesia inhalation induction
  Groups: Paediatric patients with inhalation induction
Procedure: Intravenous induction — For the intravenous induction, commonly used induction anaesthetics will be used (propofol, etomidate, ketamine, midazolam).
  Other Names: Anaesthesia intravenous induction
  Groups: Paediatric patients with intravenous induction

SUMMARY:
Intravenous anaesthesia induction is nowadays considered as gold standard, mainly because of the possibility of the rapid therapeutic intervention while having secured i.v. line.

In the paediatric patients, apart from intravenous induction, it is also possible to use in the specific situations inhalation anaesthesia induction with sevoflurane (in the mixture with O2 + air, or O2 + N2O) and secure the i.v. line afterwards in the inhalation anaesthesia. This method is in the paediatric population currently preferred, mainly because of possible fear of the painful venipuncture.

Inhalation anaesthesia induction is possible only in patients without the risk of aspiration/regurgitation of stomach content and in patients without predicted difficult airway. Even if sedative premedication is used, during the inhalation induction excitation stage of the general anaesthesia variably appears, during which hemodynamic sympathoadrenal response and involuntary limbs movement might occur. When deepening inhalation anaesthesia, progression to surgical stage and automatic breathing onset appears. This subsequently facilitates to secure the venous access, without which is is not possible to secure the airway (in exception of the emergency situations - resuscitation).

DETAILED DESCRIPTION:
The aim of this prospective observational trial is to compare the duration of inhalation and intravenous anaesthesia induction in paediatric patients, who undergo elective surgical or diagnostic procedures. After the approval of the study by the Ethics Committee of the University hospital Brno and registration of the protocol at clinicaltrials.gov, the duration of inhalation and intravenous anaesthesia induction in the patients undergoing general anaesthesia in the Departement of paediatric anaesthesia and intensive care unit, University Hospital Brno in the term from 1.9.2020 until 30.6.2021 will be measured. Measurement will be done in all patients in the given time period, who will undergo elective surgical or diagnostic procedure. The measurement will begin after the patient's arrival at the operating theatre, after the control of the documentation and beginning of the vital signs monitoring. The measurement will be terminated at the occurence of the first end-tidal carbon dioxide (ETCO2) wave, after securing the airway with laryngeal mask or orotracheal intubation

For the inhalation induction sevoflurane will be used (in the mixture with O2 + air, or O2 + N2O), for the intravenous induction, commonly used induction anaesthetics will be used (propofol, etomidate, ketamine, midazolam).

The type and the dose of the induction anaesthetic agent will be recorded (in the case of inhalation induction the dose of inhalation anaesthetic set on the vaporizer, in the case of intravenous induction the dose in mg/kg body weight).

The type and dose of the sedative premedication will be recorded, the number of attempts needed to secure i.v. line, success rate of securing the i.v. line while using Eutectic Mixture of Local Anesthetics (EMLA) patch and/or Buzzy (vibration device for patient distraction), the number of attempts needed to secure the airway, incidence of adverse events which might occur during anaesthesia induction (tachycardia, bradycardia, bronchospasm, laryngospasm).

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients scheduled for elective surgical or diagnostic procedure in the term from 10.9.2020 until 30.6.2021.

Exclusion Criteria:

* Patients in the age from 0 to 1 month
* patients with predicted difficult airway
* emergency/urgent surgeries
* patients at the risk of regurgitation/aspiration of the stomach content
* procedures in which the airway will not be secured with laryngeal mask or orotracheal intubation
* cases were the time of induction can not be measured
* patients with intravenous line in situ

Ages: 28 Days to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients scheduled for elective surgical or diagnostic procedure in the term from 10.9.2020 until 30.6.2021.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
duration of anaesthesia induction | Intraoperatively
  The average duration of inhalation and intravenous anaesthesia induction will be measured, defined as the time since the beginning of monitoring of the vital functions (ECG, pulse oximetry, non-invasive blood pressure measurement) until the first ETCO2 wave.

SECONDARY OUTCOMES:
The number of attempts needed to secure i.v. line | Intraoperatively
  The number of attempts needed to secure i.v. line will be measured
success rate of securing the i.v. line while using EMLA patch and/or Buzzy | Intraoperatively
  success rate of securing the i.v. line while using EMLA patch and/or Buzzy will be measured
Airway management | Intraoperatively
  The number of attempts needed to secure the airway will be measured
incidence of adverse events | Intraoperatively
  incidence of adverse events which might occur during anaesthesia induction (tachycardia, bradycardia, bronchospasm, laryngospasm)
Type of premedication | Intraoperatively
  type of the sedative premedication
Dose of premedication | Intraoperatively
  dose of the sedative premedication

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof. MD., Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided